CLINICAL TRIAL: NCT05581615
Title: Randomized Four-arm Trial Investigating the Effects of Different Food Matrices on the Prebiotic Efficacy of Inulin Type Fructans (ITF) From Chicory Root
Brief Title: Influence of Food Matrix on Prebiotic Efficacy in Inulin Type Fructans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY Number - 36/2020
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: gut microbiota, prebiotic intake, Bifidobacterium
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pure inulin (Active Comparator): 2 x 5 g/d inulin
  Interventions: Other: Inulin
- Shortbread containing inulin (Experimental): 2 x per day shortbread containing 5 g inulin per serving
  Interventions: Other: Inulin
- Rice drink containing inulin (Experimental): 2 x per day rice drink containing 5 g inulin per serving
  Interventions: Other: Inulin
- Milk chocolate containing inulin (Experimental): 2 x per day milk chocolate containing 5 g inulin per serving
  Interventions: Other: Inulin

INTERVENTIONS:
Other: Inulin — Each intervention provided 10 g/d inulin split into two dosages of 5 g.

SUMMARY:
The aim of the study is to investigate whether the food matrix has an influence on the prebiotic efficacy (bifidobacteria growth) of chicory-derived Orafti® inulin in healthy adult volunteers. The main question it aims to answer is:

Does the food matrix influence the prebiotic effect of chicory-derived inulin in terms of stimulation of bifidobacteria in the gut microbiota Participants will receive one of three food items containing inulin or pure inulin dissolved in water daily for 10 days. The food items or pure inulin powder will deliver 10 g/d inulin split into two dosages of 5 g/d. They will provide stool samples before and at the end of the intake period. They will record any gastrointestinal sensations and bowel habits in a diary. Urinary samples will be collected at baseline and end of intervention for analysis of metabolites with Nuclear Magnetic resonance (NMR).

ELIGIBILITY:
Inclusion Criteria:

* Volunteer is healthy at the time of pre-examination
* Volunteer is aged ≥ 18 to ≤ 65 years at the time of pre-examination
* Volunteer's BMI is ≥ 18,5 and ≤ 29,9
* Volunteer follows an average Western European diet
* Volunteer has a stool frequency of at least 3 bowel movements per week
* Volunteer is able and willing to comply with the study instructions
* Volunteer is suitable for participation in the study according to the investigator/study personnel
* Written informed consent is given by volunteer

Exclusion Criteria:

* No command of any local language
* Gastrointestinal disorders including irritable bowel syndrome (IBS), inflammatory bowel disease (IBD) or other conditions that might affect the gut environment
* Food allergies or intolerances
* Vegetarians, vegans and/or extreme diets including high protein/fibre, ketogenic, intermittent fasting and/or carnivore
* Using drugs (e.g. antibiotics, aspirin, proton pump inhibitors) influencing gastrointestinal function (8 weeks before intervention)
* Use of laxatives and labelled pre- and probiotics in the previous 4 weeks before the beginning of intervention
* Clinically significant diabetes
* Volunteers currently involved or will be involved in another clinical or food study
* History of drug (pharmaceutical or recreational) or alcohol abuse.
* Has received bowel preparation for investigative procedures in the 4 weeks prior to the study
* Has undergone surgical resection of any part of the bowel.
* If participants are pregnant or are lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Changes in level of Bifidobacterium spp. | 10 days
  Bifidobacterium spp. will be assessed by fluorescence in situ hybridisation - flow cytometry (FISH-FLOW) and 16S rRNA gene sequencing

SECONDARY OUTCOMES:
Changes in level of total Bacteria | 10 days
  Total bacteria will be assessed by fluorescence in situ hybridisation - flow cytometry (FISH-FLOW)
Changes in gut bacterial composition | 10 days
  Bacterial numbers will be assessed by fluorescence in situ hybridisation - flow cytometry (FISH-FLOW) and 16S rRNA gene sequencing
Stool frequency | 10 days
  Numbers of stools will be recorded in daily diary
Stool consistency | 10 days
  Stool consistency will be recorded in daily diary according to Bristol Stool Form Scale
Bloating | 10 days
  Bloating will be recorded in daily diary according to a 4-point scale
Abdominal pressure | 10 days
  Abdominal pressure will be recorded in daily diary according to a 4-point scale
Abdominal pain | 10 days
  Abdominal pain will be recorded in daily diary according to a 4-point scale
Flatulence | 10 days
  Flatulence will be recorded in daily diary according to a 4-point scale
Changes in urinary metabolites | 10 days
  Urinary metabolites will be analysed by Nuclear magnetic resonance (NMR)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Rastall, Prof, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No